CLINICAL TRIAL: NCT03504241
Title: Donor-derived Mesenchymal Stromal Cells, Alemtuzumab, Co-stimulation Blockade and Sirolimus for Tolerance Induction in Adult Kidney Allograft Recipients (ITN062ST)
Brief Title: Tolerance by Engaging Antigen During Cellular Homeostasis
Acronym: TEACH
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN062ST; UM1AI109565 (NIH); NIAID CRMS ID#: 20676 (Other: DAIT NIAID)
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplantation; Renal Transplantation; Renal Transplant Recipient
Keywords: mesenchymal stromal cells (MSCs); anti-rejection drugs; operational tolerance
MeSH Terms: interventions — Alemtuzumab; Abatacept; Sirolimus; Mycophenolic Acid; Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MSCs 10^4 cells/kg+anti-rejection drugs (Experimental): The first dosing cohort of 2 participants will receive 12 infusions of 10^4 donor-derived Mesenchymal Stromal Cells (MSCs) cells/kg every 4-weeks.
  Interventions: Biological: Donor-derived Mesenchymal Stromal Cells; Drug: alemtuzumab; Drug: belatacept; Drug: sirolimus; Drug: mycophenolate mofetil; Drug: mycophenolate acid; Drug: prednisone
- MSCs 10^5 cells/kg+anti-rejection drugs (Experimental): If the first 3 infusions of 10^4 donor-derived Mesenchymal Stromal Cells (MSCs) cells/kg are well tolerated, this cohort of 2 participants will receive 12 infusions of 10^5 cells/kg every 4-weeks.
  Interventions: Biological: Donor-derived Mesenchymal Stromal Cells; Drug: alemtuzumab; Drug: belatacept; Drug: sirolimus; Drug: mycophenolate mofetil; Drug: mycophenolate acid; Drug: prednisone

INTERVENTIONS:
Biological: Donor-derived Mesenchymal Stromal Cells — These MSCs are a cellular product derived from bone marrow and propagated ex vivo using FDA-approved, clinically applicable methods. Their use in kidney transplantation has been associated with a good safety profile.
  Other Names: Donor-derived MSCs; human bone marrow derived MSCs; hBM-MSC; EPIC-MSC-ITN2015-IVF-0X
Drug: alemtuzumab — Alemtuzumab, 30 mg, given once intravenously (IV) over three hours. The infusion of alemtuzumab shall begin within 24 hours of transplantation surgery and shall be given prior to the first dose of belatacept.
  Other Names: Campath®; Lemtrada®
Drug: belatacept — Belatacept will be given as an intravenous (IV) infusion of 10mg /kg over 1 hour on transplantation postoperative Day 0, Days 5 and 14, then every 2 weeks (± 2 days) for 5 additional doses.Thereafter, belatacept will be given once every 4 weeks (± 5 days) at 10 mg/kg through 24 weeks post-transplant, then at 5 mg/kg every 4-weeks until the participant is evaluated for belatacept discontinuation.
  Other Names: Nulojix®; LEA29Y
Drug: sirolimus — Rapamune® (sirolimus) (Wyeth Pharmaceuticals Inc., Philadelphia, PA) will be started on transplantation postoperative day 1 at a dose of 2 mg/day orally and adjusted to maintain goal 24-hour trough levels of 8-10 ng/ml. Participants who experience grade 3 sirolimus toxicity will undergo dose reduction.
  Other Names: Rapamune®
Drug: mycophenolate mofetil — Per protocol, and, only permitted in cases of sirolimus intolerance.
  Other Names: CellCept®
Drug: mycophenolate acid — Per protocol, and, only permitted in cases of sirolimus intolerance.
  Other Names: Myfortic®
Drug: prednisone — Per protocol, and, only permitted in cases of sirolimus intolerance.
  Other Names: corticosteroid

SUMMARY:
Anti-rejection medicines, also known as immunosuppressive drugs, are prescribed to organ transplant recipients to prevent rejection of the new organ. Long-term use of these medicines places transplant recipients at higher risk of serious infections and certain types of cancer.

The purpose of this study is to determine if:

* it is safe to give mesenchymal stromal cells (MSCs) to kidney transplant recipients, and
* the combination of the immunosuppressive (anti-rejection) study drugs plus the MSCs can allow a kidney transplant recipient to slowly reduce and/or then completely stop all anti-rejection drugs, without rejection of their kidney (renal) allograft, a process called "immunosuppression withdrawal".

DETAILED DESCRIPTION:
Background:The most common problem following a kidney transplant is the development of acute or chronic rejection. Rejection is the immunologic reaction in which the body refuses to accept the transplanted organ. The body's immune system will make destructive antibodies that will attempt to attack the transplanted organ.

In order to prevent organ rejection, all patients receiving an allograft (a graft transplanted between genetically non-identical individuals of the same species) must take anti-rejection (immunosuppressive) therapy. These medications function by lowering the body's natural immune system. Often these medications are associated with significant side effects ranging from infections to cancer.

Study:

This is a single center, open label, dose-escalation clinical trial in 6 adult recipients of Human Leukocyte Antigen (HLA)- non-identical, living-donor renal allografts. All participants will receive induction therapy with alemtuzumab followed by maintenance therapy with sirolimus and belatacept.

A total of 2 dosing cohorts of 2 recipients each will receive 12 infusions of donor-derived MSCs starting on Day 42 post-transplant and every 4 weeks starting on Day 56 post-transplant, with a minimum of 7 days between the first and second MSC infusions.

The primary objective is to determine whether immune reconstitution after lymphocyte depletion in the setting of co-stimulatory blockade and systemic MSC-derived donor antigen can promote operational tolerance in recipients of kidney allografts.

Participants will be evaluated for eligibility for sirolimus withdrawal any time between week 52 and week 104 post-transplant. Participants who successfully complete sirolimus withdrawal will remain on belatacept monotherapy for at least 24 weeks before being assessed for eligibility to discontinue belatacept. Participants who successfully complete Immunosuppression Withdrawal (ISW) will then undergo 24 weeks of high frequency follow up followed by 132 weeks of standard follow up.

Study participation may continue for up to seven (7) years after kidney transplant surgery.

*** IMPORTANT NOTICE: *** The National Institute of Allergy and Infectious Diseases and the Immune Tolerance Network do not recommend the discontinuation of immunosuppressive therapy for recipients of cell, organ, or tissue transplants outside of physician-directed, controlled clinical studies. Discontinuation of prescribed immunosuppressive therapy can result in serious health consequences and should only be performed in certain rare circumstances, upon the recommendation and with the guidance of your health care provider.

ELIGIBILITY:
Inclusion Criteria:

Recipient:

* Adult candidates of an human leukocyte antigen (HLA)-non-identical, living-donor kidney transplant:

  --Candidates must meet the United Network for Organ Sharing (UNOS) criteria, including laboratory criteria, for transplant listing;
* Evidence of established immunity to Epstein-Barr Virus (EBV) as demonstrated by serologic testing;
* Serological evidence of prior Cytomegalovirus (CMV) infection if donor is CMV positive;
* For women of child bearing potential:

  * A negative serum or urine pregnancy test with sensitivity of less than 50 mIU/mL within 72 hours of start of study medication; and
  * Agreement to use contraception:

    --- According to the FDA Office of Women's Health (http://www.fda.gov/birthcontrol), there are a number of birth control methods that are more than 80% effective

    ----Female recipients of child-bearing potential must consult with their physician and determine the most suitable method(s) from this list to be used for 18 months after the first dose of study therapy.

Donor:

* Meets institutional selection criteria for organ and bone marrow donation:

  --All donors will be screened and tested in accordance with:
  * (i) FDA 21 CRF 1271.85 requirements for donors of human cells, tissues, and cellular- and tissue-based products (HCT/P); and
  * (ii) standards for living kidney donors testing for infection established by the United Network for Organ Sharing (UNOS).
* Ability to understand and provide informed consent for all study procedures including kidney transplant and bone marrow harvest.

Exclusion Criteria:

Recipient:

* History of any immunodeficiency syndrome (including Human Immunodeficiency Virus-1 (HIV-1) and HIV-2);
* Positive anti-Hepatitis C Virus (HCV) Polymerase Chain Reaction (PCR), anti-Hepatitis C Virus (HBV) PCR, or HBV surface antigen;
* History of malignancy within 5 years of enrollment or any history of hematogenous malignancy or lymphoma; --Exception: Participants with curatively treated non-melanomatous skin cancer or curatively treated cervical carcinoma in situ may be enrolled.
* Underlying renal disease with high likelihood of recurrence, including but not limited to:

  * primary focal segmental glomerulosclerosis (FSGS),
  * Type I or II membranoproliferative glomerulonephritis (MPGN),
  * hemolytic-uremic syndrome and
  * thrombotic thrombocytopenic purpura (HUS/TTP) syndrome. ---Subject(s) with end-stage renal disease (ESRD) of unknown etiology and/or has no histologically confirmed diagnosis, may be enrolled into the study as long as there are no clinical signs or symptoms consistent with excluded clinical diagnoses.
* History of active M. tuberculosis:

  --Participants with a history of latent M. tuberculosis (LTB) as defined by positive testing for tuberculosis using an approved IGRA blood test, such as QuantiFERON®-Gold TB or T-SPOT-TB assay must:
  * have completed treatment for LTB and
  * have a negative chest x-ray. ----All participants will undergo IGRA testing for M tuberculosis within 3 months prior to transplant.
* Current or historical evidence of donor-specific antibody;
* Immunosuppressive drug therapy within one year prior to enrollment.
* May not be taking or have taken prednisone, cyclosporine A, tacrolimus, azathioprine, Mycophenolate Mofetil (MMF), cyclophosphamide, methotrexate, infliximab, etanercept, or other agents which have a primary therapeutic effect of immunosuppression in the year prior to transplantation.
* May not have taken depletional anti-lymphocyte agents at any time.

  ---Exceptions:
  * Short (≤ 30 days) courses of topical or inhaled steroids are permitted, as are
  * Short oral or parental pulses for a documented hypersensitivity reaction.
* Active autoimmune disease requiring ongoing immunosuppressive therapy or other conditions in which there is an anticipated need for immunosuppressive maintenance therapy;
* Uncompensated congestive heart failure, pulmonary edema, or symptomatic pulmonary hypertension;
* Active severe infection within a month of the screening visit;
* Use of an investigational drug within 30 days of the screening visit;
* Presence of any medical condition that the investigator deems incompatible with trial participation; or
* Inability or unwillingness to comply with protocol monitoring and therapy.

Donor:

* History of blood donation to the recipient;
* Evidence of prior Cytomegalovirus (CMV) infection if the recipient is CMV negative;
* History of HIV-1/HIV-2 infection;
* Positive HCV PCR, HBV PCR or HBV surface antigen;or
* Presence of any medical condition that the investigator deems incompatible with trial participation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who Achieve Operational Tolerance | 52 weeks after completion of Immunosuppression Withdrawal (ISW)
  Operational tolerance (to their kidney transplant) defined by participant remaining off all immunosuppression for 52 weeks after completion of Immunosuppression Withdrawal (ISW) with:
  * No evidence of biopsy-proven allograft rejection after initiation of ISW;
  * Acceptable renal function, defined as an estimated GFR > 60 ml/min/1.73cm^2 calculated using the CKD-EPI equation or a serum creatinine that has increased no more than 25% above baseline, as assessed at the week 52 visit after completion of ISW;
  * No evidence of sustained transplant renal derived pathologic proteinuria, defined as a persistent protein creatinine ratio of greater than 0.5; and
  * No Donor Specific Antibodies (DSA) at any time after completion of ISW.

SECONDARY OUTCOMES:
Proportion of Participants who Remain Off Immunosuppression | From ISW completion to end of study participation (up to approximately 5 years)
  For the duration of their study participation, after completion of immunosuppression withdrawal (ISW).
Proportion of Participants who Return to Immunosuppression | From ISW completion to end of study participation (up to approximately 5 years)
  Resumption of immunosuppressive therapy post completion of Immunosuppression Withdrawal (ISW), per standard of care.
Proportion of Participants who Achieve Belatacept Monotherapy | 48 weeks from the time of last sirolimus dose
  Belatacept monotherapy, defined as remaining on belatacept as the sole maintenance regimen for 48 weeks with:
  * No evidence of biopsy-proven allograft rejection, while on belatacept monotherapy;
  * Acceptable renal function, defined as an estimated GFR > 60 ml/min/1.73m^2 calculated using the CKD-EPI equation or a serum creatinine that has increased no more than 25% above baseline, as assessed at week 48 on belatacept monotherapy;
  * No evidence of sustained transplant renal derived pathologic proteinuria, defined as a persistent protein creatinine ratio of greater than 0.5, while on belatacept monotherapy; and
  * No Donor Specific Antibodies (DSA) at any time while on belatacept monotherapy.
Proportion of Participants who Die | From kidney transplant with alemtuzumab induction to to completion of study (up to approximately 6.5 years)
  This analysis will include all participants who provide informed consent for study participation and receive any form of study therapy including alemtuzumab, sirolimus, belatacept, or MSC infusions.
Time from Transplant to the First Episode of Rejection | From kidney transplantation to completion of study (up to approximately 7 years)
  Kaplan-Meier Analysis of time-to-occurrence to the first episode of kidney allograft rejection.
Incidence of Participants who Develop Donor Specific Antibody (DSA) | From study enrollment to completion of study (up to approximately 7 years)
  Participants that Develop de novo Anti-Human Leukocyte Antigen (HLA) Antibody or Donor Specific Antibodies (DSA).
Incidence of Adverse Events Attributable to Mesenchymal Stromal Cells (MSC) Administration | From initial MCS infusion (day 42 post kidney transplant) to end of study participation (up to 7 years)
  According to medical assessment/outcomes, investigator's brochure for MSCs, literature et al.
Frequency of Select Adverse Events (AEs) | From kidney transplantation to completion of study (up to approximately 7 years)
  Select AEs include:
  * Infection
  * Malignancy
  * Wound complications, defined as wound dehiscence, hernia or lymphocele
Incidence of Post-Transplant Diabetes | From post kidney transplantation to completion of study (up to approximately 7 years)
  New onset diabetes status post transplant (posttransplantation diabetes mellitus [PTDM])
Frequency of Antibody-Mediated Acute Cellular Rejection | From kidney transplant to completion of study (up to approximately 7 years)
  Using the 2017 Banff Classification of Renal Allograft Pathology.
Frequency of Antibody-Mediated Chronic Rejection | From kidney transplant to completion of study (up to approximately 7 years)
  Using the 2017 Banff Classification of Renal Allograft Pathology.
  As measured by the incidence of biopsy-proven chronic allograft nephropathy/IF/TA

CONTACTS AND LOCATIONS:
Overall Officials: Allan D. Kirk, M.D., Ph.D., Study Chair — Duke University Medical Center: Transplantation
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: The aim is to share data available to the public within 24 months upon completion of the study.
Access Criteria: ImmPort public data access.
URL: http://www.immport.org/immport-open/public/home/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org/
- See also: ITN's website for the study — http://www.teachstudy.org/